CLINICAL TRIAL: NCT02723058
Title: The Integrated Care Model for Homeless Mothers
Acronym: ICMHM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Linda Weinreb, Vice chair and professor, Family Medicine and Community Health, University of Massachusetts, Worcester
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34MH085881 (NIH); 1R34MH085881 (NIH)
Record Dates: First submitted 2016-03-21; First posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Depression
Keywords: Depression; Homelessness; Primary care
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICMHM (Experimental): ICMHM mothers receive services of a primary care clinician (PCP) and a care manager both trained in depression care management in a shelter-based primary care clinic.
  Interventions: Behavioral: ICMHM
- Treatment as Usual (No Intervention): Treatment as Usual mothers receive usual services of a PCP and case manager from a shelter-based primary care clinic. .

INTERVENTIONS:
Behavioral: ICMHM — ICMHM participants receive a collaborative care model adapted to include an engagement interview, attention to co-morbid conditions, and attention to basic needs.
  Arms: ICMHM

SUMMARY:
The purpose of this study is to pilot test an adapted collaborative care model for homeless mothers with depression.

DETAILED DESCRIPTION:
Homeless mothers are more vulnerable to Major Depressive Disorder (MDD) than comparable groups of impoverished mothers, with rates in recent community studies approaching 50%. Even though primary care offers an ideal venue to identify and manage depression among women who commonly fail to receive needed mental health services, rigorously tested primary care-based treatment strategies that address the needs of homeless mothers with depression are lacking. This study reports results on a pilot test and feasibility findings of a new intervention, the Integrated Care Model for Homeless Mothers (ICMHM), adapted from the collaborative care model for depression (CCM) to address unique aspects of care for homeless mothers who screened positive for depression during a shelter-based primary care visit.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who are residing in emergency shelter
* 18 years of age or older
* Screen positive for depression
* Speak English or Spanish

Exclusion Criteria:

* Not pregnant
* Not currently receiving depression treatment
* Not currently psychotic

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-12; Primary Completion 2012-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in The Hopkins Depression Symptom Checklist -Depression Scale 20 (Williams et al, 2004) | The primary end point is 6 months

SECONDARY OUTCOMES:
Number of visits to the care manager and primary care physician | The primary end point is 6 months
  Visits documented between study entry and six months recorded from EMR
New antidepressant medication prescriptions | The primary end point is 6 months
  Documentation of new antidepressant medication prescriptions between study entry and six months recorded in EMR
Patient Reactions Assessment (Galassi et al, 1992) | The primary end point is 6 months
Helping Alliance Questionnaire (Luborsky et al, 1985) | The primary end point is 6 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weinreb L, Upshur CC, Fletcher-Blake D, Reed G, Frisard C. Managing Depression Among Homeless Mothers: Pilot Testing an Adapted Collaborative Care Intervention. Prim Care Companion CNS Disord. 2016 Apr 21;18(2):10.4088/PCC.15m01907. doi: 10.4088/PCC.15m01907. eCollection 2016. PMID 27486545